CLINICAL TRIAL: NCT00954850
Title: A National Program for Severe Asthma: The Canadian Severe Asthma Network
Acronym: CSAN
Status: Withdrawn | Type: Observational
Why Stopped: Subjects not entered into electronic database due to current construct of database and associated privacy legislations within Alberta.
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Dilini Vethanayagam, Associate Professor, Medicine (Pulmonary), University of Alberta
Other Study IDs: CSAN Protocol
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2012-08-24 (Estimated); Status verified 2012-08

CONDITIONS: Severe Persistent Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — If consented to by the patient, extra clinical specimens - sputum plugs, sputum supernatant, blood and urine will be stored. If patients undergo a clinical bronchoscopy, mucosal biopsies x 2 and bronchoalveolar lavage will be stored.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Severe asthmatics: Main study group
- Mild-moderate asthmatics: Control group

SUMMARY:
The Canadian Severe Asthma Network (CSAN) was developed to gain a better understanding of the clinical, environmental, socio-economic, work-related, and biological characteristics of severe asthmatics (SA) that may account for poor response to clinically available therapies for asthma.

This network of clinical and basic researchers will be a means by which Canadian investigators can develop and conduct research in this small patient group, which could lead to better clinical management of SA.

Patient information will be entered into the CSAN database (created by PI Dr. Vethanayagam in connection with Mr. Jack Yeung) and will help researchers and doctors from multiple hospitals and universities across Canada to understand this subpopulation of asthmatics better. It will help to answer questions regarding SA epidemiology, asthma education, inflammatory monitoring, risks of near fatal asthma (NFA), symptom perception, changes in lung structure and function, co-morbidities, and the effectiveness of developing regional severe asthma clinics. Two of the early projects the investigators will be working on are psychosocial co-morbidities in asthma and medication coverage related to asthma.

There will also be biobanking of sputum samples and/or bronchoscopy samples (such as BALs & lung washings) that are being obtained for clinical purposes. Also, for those consented for biobanking blood and urine will be collected, separate from clinical care, and stored in the biobank. The Canadian Biosample Repository (CBSR) will be storing our biobanked samples. The investigators will be following the CBSR policies for storage and security. Tissue research will be conducted in the future, and separate ethics approval will be obtained for each project.

DETAILED DESCRIPTION:
5-10% of adult asthmatics have difficult to control asthma or severe asthma (SA), some of whom require systemic steroids to control their disease ("steroid dependent asthmatics"). Very little is understood about this population (Chanez, et al. JACI June 07)

Networks to study severe asthma have emerged in Europe (ENFUMOSA) and the United States (US Severe Asthma Research Program) to understand this small group of patients who account for the majority of costs related to asthma care (>50%). We would like to establish a network in Canada of well characterized asthmatics with severe asthma (and mild-moderate asthmatics as controls).

Sputum cell counts assist somewhat in improving asthma management in this population but outside of eosinophilic inflammation (one subtype) do not predict asthma control (Lemiere C et al. J Allergy Clin Immunol 2006;118:1033-9).

Little is understood regarding the many patients who do not have frequent exacerbations but rather have chronic persistent asthma (symptoms multiple times a day) particularly when non-eosinophilic. SCCs are not as useful within this group and more detailed analysis of sputum (particularly supernatant) and more invasive testing is required as we see more of this population, to better treat them.

Even less is understood about severe asthma in childhood.

We have been reviewing a few of the patients' biopsies for clues to how we can better manage them within clinical setting and note significant differences between individuals in relation to muscle mass, neuronal hypertrophy, and inflammation (which more often than not is absent in those with severe asthma).

Bronchoscopies are done routinely in SA patients to assess their airways better and obtain bronchoalveolar lavage (BAL) specimens and sometimes transbronchial biopsies.

Our hypotheses and/ or research questions are:

Immediate:

1. Natural History:

   1. What is the natural history of SA?
   2. What proportion of patients with SA and MMA have had a prior NFA episode? (retrospective)
   3. Do deaths due to asthma occur more commonly in Canadians with SA, as opposed to those with MMA? (prospective)
2. NFA and SA:

   1. What is the regional prevalence of NFA episodes in individuals with SA managed within a Canadian Health Care System?
   2. What is the natural history of patients with SA who have experienced an episode of NFA?
   3. Does management of SA within SA Centres of Excellence (SA Centres) alter the risk of subsequent episodes of NFA?
   4. What genes are related to NFA in individuals with SA and MMA?
3. What is the burden of co-morbidities in individuals with SA as opposed to individuals with MMA?
4. What is the burden of steroid-related complications in patients with SA?
5. Immunology:

   1. What is the regional prevalence of atopy in SA?
   2. What is the regional prevalence of non-TH2 mediated immunologic deviances in SA?

   Future Projects once CSAN registry is established (with specific grant funding requests)
6. Education:

   1. What are the unique educational needs of patients with SA that need to be resolved?
   2. Can we use the same translatable SA action plan in each SA Centre?
7. Inflammatory monitoring:

   1. What are the barriers to implementing the use of sputum cell counts (SCCs) routinely within SA Centres in Canada from a cost-benefit perspective?
   2. What are the barriers to establishing a standard protocol for SCC monitoring (frequency every 3 months) in SA Centres?
   3. Is there a role for Exhaled Nitric Oxide (ENO) measurement over and above SCC monitoring in SA Centres for individuals with SA?
8. Symptom perception:

   1. How does the perception of dyspnea vary in patients with NFA and those with SA?
   2. Are there simple ways to identify patients with poor perception of dyspnea in this high risk population?
9. Pathophysiology:

   1. What factors promote fixed airflow obstruction in this population?
   2. What are the features that lead to persistent airway neutrophilia in this population?
   3. Do those with SA develop more airway remodelling than those with MMA and when present, does airway remodelling progress at a faster rate in the SA group?
10. Health Service Delivery:

    1. Are there differences in organizational clinic structure of SA Centres that improve efficiency of management?
    2. Can we develop further specialized new SA Centres in Canada effectively (knowledge transfer for organization)?
    3. Is it cost effective to develop regional SA Centres in Canada?

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 and older) with physiologically confirmed SA or mild-moderate asthma and followed by an asthma specialist for at least 6 months.
* Must agree to have regular clinic visits (minimum 3-4 per year for SA, 1-2 for mild-moderate asthma).
* Must have good compliance with medications Patients with asthma and COPD.

Exclusion Criteria:

* Malignancy and other significant medical conditions that will impact follow up within this program.
* Those less than 18 years of age.
* Concomitant interstitial lung disease, sarcoidosis, other significant lung disease.
* Those who have had a transplant.
* Significant travel with work.
* Unable to make appointments (every three to six months over 2 years).
* Those residing in another country or planned absence for more than one month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe asthmatics as the primary study group, mild-moderate asthmatics as the control group
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dilini Vethanayagam, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- See also: CSAN Page — http://www.severeasthma.ca